CLINICAL TRIAL: NCT00669604
Title: Counseling on Formula Feeding and Antiretroviral Prophylaxis Successfully Reduced Transmission of HIV-1 From Mother to Child in Northern Vietnam
Brief Title: HIV Vertical Transmission in Vietnam
Status: Completed | Type: Observational
Sponsor: National Institute of Hygiene and Epidemiology, Vietnam (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Phung Dac Cam, National Institute of Hygiene and Epidemiology
Other Study IDs: 3RF-1; 3RF-1/MoST-Sida
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: HIV Infections
Keywords: Mother to child transmission of HIV; HIV infected children
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral EDTA blood samples were collected from the child at birth (1-2 days), at 1, 3, 6, 12, and 18 months of age and processed at the Molecular Laboratory in the Hanoi Obstetric and Gynaecology hospital. The maternal blood samples were taken at the same day as the first sample of their child. Three ml EDTA blood was taken from the mother and 2 ml from the child. The blood was processed within 8 hours. Cells and plasma were stored separately at - 20 Celcius degree.
Oversight: Data Monitoring Committee: No

SUMMARY:
Prevention of HIV-1 transmission from mother-to-child by non-breast-feeding is complicated by increased infant mortality in developing countries. However, extensive counselling about formula feeding turned out safe in Vietnam, a middle-income country.Extensive counselling together with formula feeding and antiretroviral therapy reduced vertical transmission of HIV-1 considerably.

DETAILED DESCRIPTION:
Observation 135 HIV mother to check up and delivery in the Obstetric and Gynecology in two big city in Northern Vietnam (Hanoi and Haiphong)and follow up their children from the birth to 18 months. They were provide the antiretroviral by the National program for prevention of mother-to-child transmission of HIV, also the counseling estimates 6 hours for each mother-child pair while study progressing. Using the Nested PCR to diagnosis HIV infected in the children in difference time point before 18 months. Our Outcome are

* The rate of HIV transmission form mother to child in our study is 6,7%(9?135). In utero is 1,5% and 5% in gestation.
* Sixty-nine percent of HIV pregnant women were get antiretroviral. Most of them (84%) get nevirapine at delivery (6 children HIV infected). The rest get triple antiretroviral(2 infected child).
* Selective cesarean section not comment for HIV pregnant women.
* Non breast feeding were recommended and all mothers chose formula feeding to their child so that we had no data for transmission by breast milk.
* Two HIV infected child die before 18months versus non die in uninfected child.
* CD4 T cell count lower than 200/microliter were observed dominate in mother infected child.

ELIGIBILITY:
Inclusion Criteria:

* HIV Mother willing to enroll to study and their child For mother: Their HIV status was diagnosed by at least one quick test and two different ELISA serological tests.

For their child: the child had tested HIV at list 3 time one at birth, one at 12 or 18 months and one in between.

Exclusion Criteria:

* The child had less than 3 time to test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-1 infected pregnant women were identified in the Obstetric and Gynaecology hospitals in Hanoi (2004-2007) and Haiphong (2006-2007).
  They were encouraged to participate in a prospective study with regular clinical follow up of their children from birth to 12-18 months of age. All participants signed an informed consent.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2004-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
HIV-infection in the children. | 2004 - 2007

SECONDARY OUTCOMES:
Mortality in the children in the first 18 months | completed 2007
Safety of formula feeding measured by the mortality by 18 months | Completed by end of 2007

CONTACTS AND LOCATIONS:
Overall Officials: Phung D Cam, MD,PhD, Study Chair — National Institute of Hygiene and Epidemiology, Vietnam
Locations (1):
- Obstetric and Gynaecology Hospital, Hanoi, Hanoi, Vietnam

REFERENCES:
- [Result] Tran Thi Thanh Ha, Pham Le Tuan, Nguyen Huy Bao et al. Successful reduction of mother-to-child transmission of HIV-1 by nevirapin and non-breastfeeding in Hanoi and Haiphong. Retrovirology 2008; 5, S1: 26-27.